CLINICAL TRIAL: NCT01933828
Title: thoracoSCopic Versus OPen Lobectomy for Early Stage Lung Cancer: a Randomized Prospective Trial
Brief Title: Treatment of Early Stage Lung Cancer by VATS Versus OPEN Lobectomy
Acronym: SCOPE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Radboud University Medical Center (Other)
Collaborators: University Medical Center Nijmegen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UMCN_NL40542.091.12
Record Dates: First submitted 2013-05-27; First posted 2013-09-02 (Estimated); Last update posted 2013-11-08 (Estimated); Status verified 2013-08

CONDITIONS: Lung Cancer
Keywords: Lung cancer; surgery video-assisted; robot; surgical treatment
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- OPEN lobectomy (Active Comparator): Lobectomy and mediastinal lymph node dissection by thoracotomy with rib-spreading.
  Interventions: Procedure: OPEN lobectomy
- VATS lobectomy (Active Comparator): Thoracoscopic minimally invasive lobectomy with thoracoscopic mediastinal lymph node dissection without rib-spreading.
  Interventions: Procedure: VATS lobectomy
- ROBOT-assisted lobectomy (Other): Robot-assisted lobectomy with mediastinal lymph node dissection (Robot group as clinical assignment in prospective Cohort).
  Interventions: Device: ROBOT-assisted lobectomy

INTERVENTIONS:
Procedure: OPEN lobectomy — Lobectomy and mediastinal lymph node dissection by thoracotomy with rib-spreading.
  Arms: OPEN lobectomy
Procedure: VATS lobectomy — Thoracoscopic minimally invasive lobectomy with thoracoscopic mediastinal lymph node dissection without rib-spreading.
  Arms: VATS lobectomy
Device: ROBOT-assisted lobectomy — Robot-assisted lobectomy with mediastinal lymph node dissection (Robot group as clinical assignment in prospective Cohort).
  Arms: ROBOT-assisted lobectomy

SUMMARY:
In patients with early stage lung cancer surgical lobectomy is the treatment of choice. A resection by Video-assisted Thoracic Surgery (VATS) is probably superior to an open procedure by thoracotomy for patients with early stage lung cancer, but randomized evidence for superiority is lacking. Furthermore, VATS lobectomy has not gained broad implementation yet. The objective of this study is to assess the benefits of VATS- over open lobectomy regarding quality of life and costs in a prospective randomized controlled multicenter trial. All patients meeting the inclusion criteria that are not randomized will be included in a prospective Cohort.

DETAILED DESCRIPTION:
Rationale: Surgical lobectomy is the treatment of choice for patients with early stage lung cancer. In some centres, video-assisted thoracic surgery (VATS) lobectomy is preferred, where other centres hold on to the conventional open lobectomy via a thoracotomy. Although several studies have demonstrated fewer postoperative complications and shorter hospital length of stay for the VATS procedure, others have reported concerns regarding oncologic equivalence, mainly based on incomplete lymph node staging. Convincing randomized evidence from the literature is lacking. The aim of this randomized multicentre study is to compare quality of life, oncologic endpoints and cost-effectiveness between VATS- and open (thoracotomy) lobectomy.

Objective: To compare quality of life, cost-effectiveness and number of dissected mediastinal lymph nodes between open,VATS and ROBOT-assisted lobectomy.

Study design: A prospective multi-centre randomized trial with a prospective registry arm Study population: Adult patients of either gender, selected by the pulmonary oncological multidisciplinary team to undergo surgical lobectomy for early-stage lung carcinoma.

Intervention: One group is assigned to the open procedure: posterolateral thoracotomy for lobectomy with mediastinal lymph node dissection. The other group is assigned to the VATS procedure: thoracoscopic minimally invasive lobectomy with thoracoscopic mediastinal lymph node dissection. All patients that do meet the inclusion criteria but are not participating in the randomized trial can be included in the prospective Cohort arm of the study evaluating clinical assignment to OPEN- VATS or ROBOT-assisted lobectomy.

Main study parameters/endpoints: Primary endpoints are postoperative quality of life, and hospital length of stay. Secondary endpoints include cancer specific quality of life, number of dissected mediastinal lymph nodes and stations, procedural complication rates, pulmonary function, overall costs and survival.

Centres participating in this study currently perform the open- and VATS and/or ROBOT-assisted lobectomy in daily clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Non-small cell lung carcinoma, pathologically confirmed or strong suspicion based on imaging.
* T1 or T2a (≤ 5 cm) on computer tomography (CT).
* Primary aim is lobectomy.
* Tumor not in close relation to the hilar structures (bronchus,vessels)based on CT.
* Clinically staged N0 (no regional lymph node metastasis) or N1 (metastasis to ipsilateral, hilar, interlobar- and/or intrapulmonary lymph nodes), M0 (no distant metastasis) after clinical staging according to the current Dutch guideline (may 2011).

Exclusion Criteria:

* T2b, T3 or T4 tumor (7th guideline TNM classification NSCLC).
* Mediastinal lymph node metastasis (N2, N3).
* Distant metastasis (M1).
* Previous thoracic surgery on same side.
* Pneumonectomy as primary aim.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 176 (Estimated)
Dates: Start 2013-06; Primary Completion 2015-06 (Estimated); Study Completion 2015-06 (Estimated)

PRIMARY OUTCOMES:
Quality of life (EQ5D) | up to12 month
  Primary endpoints include Quality of life assessed by EQ5D for VATS versus open lobectomy in patients with early stage non small cell lung carcinoma.
Hospital length of stay | day of discharge from hospital after surgery (expected within 2 weeks).

SECONDARY OUTCOMES:
cancer specific quality of life (QLQ C30 and 13) | preoperatively 1 week before surgery and at 3-6 and 12 month
number of dissected mediastinal lymphnode stations | day 0 (intraoperatively)
  The number of intraoperatively dissected mediastinal lymphnode stations is assessed as a secondary oncologic outcome measure.
composite endpoint of intra- and postoperative complications | form the day of surgery up to discharege (expected within 2 weeks)
  This secondary composite endpoints include conversion rate, bleeding, air leakage, pain, cardiac arrhythmias, wound infection, pulmonary complications, pulmonary function.

CONTACTS AND LOCATIONS:
Overall Officials: A. Verhagen, MD, Principal Investigator — Radboud University Nijmegen Medical Center, Department of Cardio-thoracic Surgery Route 677 Postbus 9101, 6500 HB Nijmegen Tel: + 31 24 361 47 44 Fax: +31 24 354 01 29; T. van Brakel, MD, PhD, Principal Investigator — Radboud University Nijmegen Medical Center, Department of Cardio-thoracic Surgery Route 677 Postbus 9101, 6500 HB Nijmegen Tel: + 31 24 361 47 44 Fax: +31 24 354 01 29
Locations (1):
- Radboud University Nijmegen Medical Center, Department of Cardio-thoracic Surgery, Nijmegen, Netherlands